CLINICAL TRIAL: NCT02154139
Title: Leuplin SR 11.25 mg for Injection Specified Drug-use Survey "Long-term Use Survey on Premenopausal Breast Cancer Patients (96 Weeks)"
Brief Title: Leuprorelin Acetate SR 11.25 mg for Injection Specified Drug-use Survey "Long-term Use Survey on Premenopausal Breast Cancer Patients (96 Weeks)"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 265-201; JapicCTI-142516 (Registry Identifier: JapicCTI); JapicCTI-R150796 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-04-23; First posted 2014-06-03 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Pharmacological therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Leuprolide; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- leuprorelin acetate: Subcutaneous administration of leuprorelin acetate once every 12 weeks
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: Leuprorelin acetate — Leuprorelin acetate SR 11.25 mg for injection
  Other Names: Leuplin SR 11.25 mg for Injection

SUMMARY:
The purpose of this survey is to examine the safety and efficacy of long-term use (96 weeks) of leuprorelin acetate SR (slow release) 11.25 milligram (mg) for injection (Leuplin SR 11.25 mg for Injection) in premenopausal breast cancer patients in daily medical practice, as well as to examine factors that can influence the safety and efficacy of treatment with leuprorelin acetate SR 11.25 mg for injection (Leuplin SR 11.25 mg for Injection).

DETAILED DESCRIPTION:
This survey was designed to examine the safety and efficacy of long-term use (96 weeks) of leuprorelin acetate 3 months depot for injection (Leuplin SR 11.25 mg for Injection) in premenopausal breast cancer patients in daily medical practice, as well as to examine factors that can influence the safety and efficacy of treatment with leuprorelin acetate SR 11.25 mg for injection (Leuplin SR 11.25 mg for Injection).

For adults, 11.25 mg of leuprorelin acetate is usually administered subcutaneously once every 12 weeks. Prior to injection, the plunger rod of the syringe is pushed upward with the needle pointed upward, allowing the entire suspension fluid contained to be transferred to the powder. The powder is then fully suspended in the fluid while ensuring that bubbles are not generated.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal breast cancer patients (patients with advanced or recurrent breast cancer and patients who received adjuvant therapy).

Exclusion Criteria:

* Patients with a history of treatment with Leuplin SR 11.25 mg for Injection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 157 investigative site in Japan from 26-Dec-05 to 31-Mar-10.
Pre-assignment Details: Participants with a historical diagnosis of premenopausal breast cancer (advanced or recurrent) who were treated with Leuprorelin Acetate 11.25 milligrams (mg) in daily medical practice along with adjuvant therapy were observed.
Groups:
- Leuprorelin Acetate: Leuprorelin Acetate 11.25 mg, injection subcutaneously once every 12 weeks up to 96 weeks.
Period: Overall Study
Arm/Group | Leuprorelin Acetate
Started | 651
Completed | 644
Not Completed | 7
Not completed — Injection not administered | 2
Not completed — Other | 2
Not completed — Investigator transferred | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as participants who were enrolled and completed the study.
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 644
Age, Customized [Number; unit: participants]
  20-29 years | 11
  30-34 years | 47
  35-39 years | 113
  40-44 years | 201
  45-49 years | 212
  50-55 years | 58
  Unknown | 2
Sex/Gender, Customized [Number; unit: participants] — Only female participants were enrolled in the study.
  participants | 644
Stage of primary lesion [Number; unit: participants] — Tumor Node Metastasis (TNM):based on tumor size, if cancer cells had spread to nearby lymph nodes (LN), or distant metastasis. Stages included: stage 0(no evidence of cancer cells),stage 1(T1N0M0), stage IIA(T0N1M0, T1N1M0, T2N0M0), stage IIB(T2N1M0, T3N0M0), stage IIIA(T0N2M0, T1N2M0, T2N3M0, T3N1orN2M0),stage IIIb( T4 anyNM0, any TN3M0),stage IIIC(any TN3M0), stage IV(any T any NM1), where T0=early form of tumor, T1=<2 centimeter (cm), T2=2-5 cm, T3=>2 cm, T4=large sized, N0=not spread to LN, N1=spread to 1 to 3,N2=spread to 4 to 9,N3=spread >10 axillary LN, M0=no metastasis, M1= Metastasis.
  participants
    T0N0M0 | 2
    Stage 0 | 17
    Stage I | 265
    Stage IIA | 199
    Stage IIB | 85
    Stage IIIA | 24
    Stage IIIB | 6
    Stage IIIC | 1
    Stage IV | 23
    Unclassifiable | 22
Recurrence prior to start of treatment with leuprorelin acetate 11.25 mg for injection [Number; unit: participants]
  Experienced recurrence | 50
  No recurrence observed | 594
Performance Status (at the start of treatment with leuprorelin acetate 11.25 mg for injection) [Number; unit: participants] — Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair.
  participants
    0 | 602
    1 | 33
    2 | 3
    3 | 4
    4 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AE) which are in the investigator's opinion of causal relationship to the study treatment. AE are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to 96 weeks
Population: Safety analysis set was defined as participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 644
participants | 128

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAE) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The event occurred was breast cancer female
Time Frame: Baseline up to 96 weeks
Population: Safety analysis set was defined as participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 644
participants | 1

3. Secondary Outcome: Percentage of Participants With Advanced or Recurrent Breast Cancer (Best Response)
Description: Best overall response for a participant is the best observed post-baseline disease response as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 criteria. Objective response was defined as a complete response (CR) or partial response (PR) determined on 2 consecutive occasions greater than or equal to (>=) 4 weeks apart, using Response Evaluation Criteria in Solid Tumors (RECIST). CR: The disappearance of all target lesions and all non-target lesions, normalization of tumor marker level, and no new lesions. PR: Disappearance of all target lesions and persistence of >= 1 non-target lesions and/or the maintenance of tumor marker level above the normal limits, or, at least a 30 percent (%) decrease in the sum of the longest diameter of target lesions, and no new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Week 24, 48,96
Population: The efficacy assessment population was defined as participants with advanced or recurrent breast cancer whose efficacy data at baseline and at least 1 post-baseline time points was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 48
percentage of participants
  Week 24 | 10.34 [2.19 to 27.35]
  Week 48 | 12.00 [2.55 to 31.22]
  Week 96 | 15.00 [3.21 to 37.89]

4. Secondary Outcome: Percentage of Participants With Progression Free Survival
Description: Progression-free survival (PFS) was defined as the time from the first day of study treatment to documented disease progression or death on study (ie, death from any cause within 30 days of the last dose of study drug), whichever occurred first. Disease progression was at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. For patients who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: Baseline up to 96 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 44
percentage of participants | 49.68 [32.47 to 64.73]

5. Secondary Outcome: Percentage of Participants With Recurrence-free Survival Who Were Treated With the Drug as Adjuvant Therapy
Description: Recurrence-free survival was determined in participants who were treated with the drug as adjuvant therapy, and tabulated, based on the date recurrence is confirmed, the presence or absence of recurrence, continued survival or death, and the date of death.
Time Frame: Baseline up to 96 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 522
percentage of participants | 95.37 [92.96 to 96.96]

ADVERSE EVENTS:
Time Frame: Baseline up to 96 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Leuprorelin Acetate
Serious Adverse Events (participants affected / at risk) | 20/644
Other Adverse Events (participants affected / at risk) | 76/644
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate (N=644)
Condition aggravated (General disorders) | 3
Pyrexia (General disorders) | 1
Blood amylase increased (Investigations) | 1
Carbohydrate antigen 15-3 increased (Investigations) | 1
Urine amylase increased (Investigations) | 1
Completed suicide (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate (N=644)
Injection site induration (General disorders) | 41
Hot flush (Vascular disorders) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.